CLINICAL TRIAL: NCT04547712
Title: Adaptive DBS Algorithm for Personalized Therapy in Parkinson's Disease (ADAPT-PD)
Brief Title: Adaptive DBS Algorithm for Personalized Therapy in Parkinson's Disease
Acronym: ADAPT-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MDT19001
Record Dates: First submitted 2020-08-20; First posted 2020-09-14 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Randomization to a crossover sequence of aDBS single threshold and aDBS dual threshold modes
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- aDBS Single Threshold (Experimental): Adaptive DBS Single Threshold Mode
  Interventions: Device: Adaptive DBS
- aDBS Dual Threshold (Experimental): Adaptive DBS Dual Threshold Mode
  Interventions: Device: Adaptive DBS

INTERVENTIONS:
Device: Adaptive DBS — Subjects for whom both aDBS modes are acceptable will receive Dual and Single Threshold aDBS
  Other Names: aDBS

SUMMARY:
The purpose of the study is to demonstrate the safety and effectiveness of adaptive DBS (aDBS) for Parkinson's disease.

DETAILED DESCRIPTION:
Prospective single-blind, randomized crossover, multi-center study of aDBS in subjects with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

General

1. Subject has idiopathic Parkinson's disease
2. Subject is implanted with Percept PC (Model B35200) and Medtronic Deep Brain Stimulation (DBS) leads (Model 3387, 3389, B33005 or B33015) and extensions (Model 37085, 37086, or B34000) bilaterally in the same target (physician confirmed), subthalamic nucleus (STN) or Globus Pallidus (GPi)
3. In the opinion of the investigator, the subject responds to DBS Therapy.
4. Based on the opinion of the investigator, the subject's cDBS parameters and PD medications are stable and expected to remain stable from enrollment through the end of the aDBS Evaluation phase
5. (Primary Cohort) Subject is configured to ring mode monopolar or dual monopolar stimulation using contacts 1 and/or 2 (9 and/or 10) on at least one side.

5. (Directional Stimulation Cohort) Subject is configured to directional monopolar or dual monopolar stimulation using contacts 1 and/or 2 (9 and/or 10) 6. Subject is willing and able to attend all study-required visits and complete the study procedures (e.g. 1-month recall questionnaires, MDS-UPDRS III) 7. Subject has the ability to understand and provide written informed consent for participation in the study prior to the study-related procedures being conducted 8. Subject is a male or non-pregnant female. If female of child-bearing potential, and if sexually active, must be using, or agree to use, a medically-acceptable method of birth control as confirmed by the investigator 9. For subjects with the SenSight system: Subject is configured to the following stimulation rates: 55, 85, 110, 125, 145, 164 or 180 Hz (as required for sensing/aDBS)

Local Field Potential (LFP) Screening Inclusion Criteria

1. Subject has required Alpha-Beta band (8-30 Hz) amplitude ≥ 1.2 µVp detected on either left and/or right DBS leads

Exclusion Criteria:

1. Subject and/or caregiver is unable to utilize the patient programmer
2. Subject has more than one lead in each hemisphere of the brain
3. Subject has cortical leads or additional unapproved hardware implanted in the brain
4. Subject has more than one INS
5. At enrollment, the subject's INS has a predicted battery life of <1 year
6. Subject has Beck Depression Inventory II (BDI-II) > 25
7. Subject requires diathermy, transcranial magnetic stimulation (TMS), or electroconvulsive therapy (ECT)
8. Subject has a metallic implant in the head, (eg, aneurysm clip, cochlear implant)
9. Subject has, or plans to obtain, an implanted electrical stimulation medical device anywhere in the body (eg, cardiac pacemaker, defibrillator, spinal cord stimulator)
10. Subject has, or plans to obtain, an implanted medication pump for the treatment of Parkinson's disease (eg, DUOPATM infusion pump) and/or portable infusion pump
11. Based on the opinion of the investigator, the subject has an abnormal neurological examination that would preclude them from study participation
12. Subject is breast feeding
13. Subject is under the age of 18 years
14. Subject is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound the results of this study as determined by the Medtronic study team
15. Subject is unable to use or tolerate wearable
16. Subjects with signal artifact on all 6 aDBS sense pathways (3 each on both DBS leads) which preclude the clinician from setting thresholds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2025-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Bronte-Stewart, MD, MSE, Principal Investigator — Stanford University
Locations (10):
- United States (7):
  - University of California San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - University of Florida, Gainesville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Toronto Western Hospital, Toronto, Ontario, Canada
- UJF Grenoble, Grenoble, France
- Amsterdam UMC, location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bronte-Stewart HM, Beudel M, Ostrem JL, Little S, Almeida L, Ramirez-Zamora A, Fasano A, Hassell T, Mitchell KT, Moro E, Gostkowski M, Chattree G, de Bie RMA, de Neeling M, Pina-Fuentes D, Swinnen B, Starr PA, Hammer LH, Foote KD, Richardson RM, Flaherty A, Boogers A, Sa'di Q, Meoni S, Castrioto A, Stanslaski S, Summers RLS, Tonder L, Tan Y, Berrier H, Goble TJ, Raike RS, Herrington TM; ADAPT-PD Investigators. Long-Term Personalized Adaptive Deep Brain Stimulation in Parkinson Disease: A Nonrandomized Clinical Trial. JAMA Neurol. 2025 Nov 1;82(11):1171-1180. doi: 10.1001/jamaneurol.2025.2781. PMID 40982287
- [Derived] Swinnen BEKS, Buijink AW, Pina-Fuentes D, de Bie RMA, Beudel M. Diving into the subcortex: The potential of chronic subcortical sensing for unravelling basal ganglia function and optimization of deep brain stimulation. Neuroimage. 2022 Jul 1;254:119147. doi: 10.1016/j.neuroimage.2022.119147. Epub 2022 Mar 27. PMID 35346837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 85 subjects were enrolled between December 14, 2020 and July 29, 2022 at 12 centers located in the US, Europe, and Canada. Out of these 85 subjects, 68 were in Primary Cohort and 17 in Directional Stimulation Cohort.
Pre-assignment Details: 60 out of 85 subjects entered into the aDBS Evaluation Phase of the study. Of those 25 who didn't enter into the aDBS Evaluation Phase, 1 had inclusion/exclusion screen failure, 12 LFP screen failures, 4 physician decisions, and 8 subject decisions.
Groups:
- Primary Cohort, Crossover Sequence 1: aDBS Single Threshold Mode, Then aDBS Dual Threshold Mode: This cohort comprised of study subjects implanted with legacy lead model 3387 or 3389, or with SenSight™ lead model B33005 or B33015 programmed to ring mode stimulation, received Single Threshold evaluation for about one month first, then Dual Threshold evaluation for about one month.
- Primary Cohort, Crossover Sequence 2: aDBS Dual Threshold Mode, Then aDBS Single Threshold Mode: This cohort comprised of study subjects implanted with legacy lead model 3387 or 3389, or with SenSight™ lead model B33005 or B33015 programmed to ring mode stimulation, received Dual Threshold evaluation for about one month first, then Single Threshold evaluation for about one month.
- Primary Cohort, One Mode: aDBS Single Threshold Mode: This cohort comprised of study subjects implanted with legacy lead model 3387 or 3389, or with SenSight™ lead model B33005 or B33015 programmed to ring mode stimulation, received only Single Threshold evaluation for about one month.
- Primary Cohort, One Mode: aDBS Dual Threshold Mode: This cohort comprised of study subjects implanted with legacy lead model 3387 or 3389, or with SenSight™ lead model B33005 or B33015 programmed to ring mode stimulation, received only Dual Threshold evaluation for about one month.
- Directional Stimulation Cohort, Crossover Sequence 1: aDBS Single, Then aDBS Dual Threshold Mode; Directional Stimulation Cohort, Crossover Sequence 2: aDBS Dual, Then aDBS Single Threshold Mode; Directional Stimulation Cohort, One Mode: aDBS Dual Threshold Mode: This cohort comprised of study subjects with SenSight™ lead model B33005 or B33015 programmed to directional stimulation, with Single and/or Dual Threshold evaluation for about one month.
Period: cDBS Baseline (~ 30 Days)
Arm/Group | Primary Cohort, Crossover Sequence 1: aDBS Single Threshold Mode, Then aDBS Dual Threshold Mode | Primary Cohort, Crossover Sequence 2: aDBS Dual Threshold Mode, Then aDBS Single Threshold Mode | Primary Cohort, One Mode: aDBS Single Threshold Mode | Primary Cohort, One Mode: aDBS Dual Threshold Mode | Directional Stimulation Cohort, Crossover Sequence 1: aDBS Single, Then aDBS Dual Threshold Mode | Directional Stimulation Cohort, Crossover Sequence 2: aDBS Dual, Then aDBS Single Threshold Mode | Directional Stimulation Cohort, One Mode: aDBS Dual Threshold Mode
Started | 16 | 14 | 5 | 10 | 6 | 7 | 2
Completed | 16 | 14 | 5 | 10 | 6 | 7 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: aDBS Setup & Adjustment (up to 65 Days)
Arm/Group | Primary Cohort, Crossover Sequence 1: aDBS Single Threshold Mode, Then aDBS Dual Threshold Mode | Primary Cohort, Crossover Sequence 2: aDBS Dual Threshold Mode, Then aDBS Single Threshold Mode | Primary Cohort, One Mode: aDBS Single Threshold Mode | Primary Cohort, One Mode: aDBS Dual Threshold Mode | Directional Stimulation Cohort, Crossover Sequence 1: aDBS Single, Then aDBS Dual Threshold Mode | Directional Stimulation Cohort, Crossover Sequence 2: aDBS Dual, Then aDBS Single Threshold Mode | Directional Stimulation Cohort, One Mode: aDBS Dual Threshold Mode
Started | 16 | 14 | 5 | 10 | 6 | 7 | 2
Completed | 16 | 14 | 5 | 10 | 6 | 7 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Crossover: 1st Intervention (~ 30 Days)
Arm/Group | Primary Cohort, Crossover Sequence 1: aDBS Single Threshold Mode, Then aDBS Dual Threshold Mode | Primary Cohort, Crossover Sequence 2: aDBS Dual Threshold Mode, Then aDBS Single Threshold Mode | Primary Cohort, One Mode: aDBS Single Threshold Mode | Primary Cohort, One Mode: aDBS Dual Threshold Mode | Directional Stimulation Cohort, Crossover Sequence 1: aDBS Single, Then aDBS Dual Threshold Mode | Directional Stimulation Cohort, Crossover Sequence 2: aDBS Dual, Then aDBS Single Threshold Mode | Directional Stimulation Cohort, One Mode: aDBS Dual Threshold Mode
Started | 16 | 14 | 0 (The flow of the participants from One Mode is addressed in the periods for One Mode.) | 0 (The flow of the participants from One Mode is addressed in the periods for One Mode.) | 6 | 7 | 0 (The flow of the participants from One Mode is addressed in the periods for One Mode.)
Completed | 16 | 14 | 0 | 0 | 6 | 7 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Crossover: 2nd Intervention (~ 30 Days)
Arm/Group | Primary Cohort, Crossover Sequence 1: aDBS Single Threshold Mode, Then aDBS Dual Threshold Mode | Primary Cohort, Crossover Sequence 2: aDBS Dual Threshold Mode, Then aDBS Single Threshold Mode | Primary Cohort, One Mode: aDBS Single Threshold Mode | Primary Cohort, One Mode: aDBS Dual Threshold Mode | Directional Stimulation Cohort, Crossover Sequence 1: aDBS Single, Then aDBS Dual Threshold Mode | Directional Stimulation Cohort, Crossover Sequence 2: aDBS Dual, Then aDBS Single Threshold Mode | Directional Stimulation Cohort, One Mode: aDBS Dual Threshold Mode
Started | 16 | 14 | 0 | 0 | 6 | 7 | 0
Completed | 16 | 14 | 0 | 0 | 6 | 7 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: One Mode: Single Threshold (~ 30 Days)
Arm/Group | Primary Cohort, Crossover Sequence 1: aDBS Single Threshold Mode, Then aDBS Dual Threshold Mode | Primary Cohort, Crossover Sequence 2: aDBS Dual Threshold Mode, Then aDBS Single Threshold Mode | Primary Cohort, One Mode: aDBS Single Threshold Mode | Primary Cohort, One Mode: aDBS Dual Threshold Mode | Directional Stimulation Cohort, Crossover Sequence 1: aDBS Single, Then aDBS Dual Threshold Mode | Directional Stimulation Cohort, Crossover Sequence 2: aDBS Dual, Then aDBS Single Threshold Mode | Directional Stimulation Cohort, One Mode: aDBS Dual Threshold Mode
Started | 0 (The flow of the participants from the Crossover arm is addressed in the periods for Crossover Sequences.) | 0 (The flow of the participants from the Crossover arm is addressed in the periods for Crossover Sequences.) | 5 (The flow of the participants from Single Threshold Mode is addressed in the period for One Mode - Single Threshold.) | 0 | 0 (The flow of the participants from the Crossover arm is addressed in the periods for Crossover Sequences.) | 0 (The flow of the participants from the Crossover arm is addressed in the periods for Crossover Sequences.) | 0
Completed | 0 | 0 | 5 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: One Mode: Dual Threshold (~ 30 Days)
Arm/Group | Primary Cohort, Crossover Sequence 1: aDBS Single Threshold Mode, Then aDBS Dual Threshold Mode | Primary Cohort, Crossover Sequence 2: aDBS Dual Threshold Mode, Then aDBS Single Threshold Mode | Primary Cohort, One Mode: aDBS Single Threshold Mode | Primary Cohort, One Mode: aDBS Dual Threshold Mode | Directional Stimulation Cohort, Crossover Sequence 1: aDBS Single, Then aDBS Dual Threshold Mode | Directional Stimulation Cohort, Crossover Sequence 2: aDBS Dual, Then aDBS Single Threshold Mode | Directional Stimulation Cohort, One Mode: aDBS Dual Threshold Mode
Started | 0 | 0 | 0 (The flow of the participants from Single Threshold Mode is addressed in the period for One Mode - Single Threshold.) | 10 (The flow of the participants from Dual Threshold Mode is addressed in the period for One Mode - Dual Threshold.) | 0 | 0 | 2 (The flow of the participants from Dual Threshold Mode is addressed in the period for One Mode - Dual Threshold.)
Completed | 0 | 0 | 0 | 10 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The 60 subjects who entered into the aDBS Evaluation Phase of the study are summarized for baseline characteristics so that arms/groups can be assigned based on the flowchart.
Groups:
- Directional Stimulation Cohort, One Mode: aDBS Dual Threshold Mode: This cohort comprised of study subjects with SenSight™ lead model B33005 or B33015 programmed to directional stimulation, with Dual Threshold evaluation for about one month.
- Total: Total of all reporting groups
Arm/Group | Primary Cohort, Crossover Sequence 1: aDBS Single Threshold Mode, Then aDBS Dual Threshold Mode | Primary Cohort, Crossover Sequence 2: aDBS Dual Threshold Mode, Then aDBS Single Threshold Mode | Primary Cohort, One Mode: aDBS Single Threshold Mode | Primary Cohort, One Mode: aDBS Dual Threshold Mode | Directional Stimulation Cohort, Crossover Sequence 1: aDBS Single, Then aDBS Dual Threshold Mode | Directional Stimulation Cohort, Crossover Sequence 2: aDBS Dual, Then aDBS Single Threshold Mode | Directional Stimulation Cohort, One Mode: aDBS Dual Threshold Mode | Total
Number analyzed (Participants) | 16 | 14 | 5 | 10 | 6 | 7 | 2 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (9.49) | 64.2 (7.62) | 59.6 (7.16) | 59.6 (10.08) | 59.7 (4.18) | 61.0 (8.08) | 58.0 (2.83) | 61.1 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 4 | 2 | 1 | 2 | 1 | 19
  Male | 12 | 9 | 1 | 8 | 5 | 5 | 1 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 13 | 10 | 2 | 7 | 5 | 6 | 2 | 45
  Unknown or Not Reported | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 13 | 11 | 2 | 5 | 4 | 6 | 2 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 3 | 3 | 1 | 1 | 0 | 14
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 4
  Netherlands | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 6
  United States | 13 | 11 | 2 | 7 | 6 | 7 | 2 | 48
  France | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of aDBS Subjects With "On" Time Without Troublesome Dyskinesia Exceeding the Threshold.
Description: In the PD Home Diary, in 30-minute intervals, patients recorded whether they were in the "On" condition (with dyskinesia, with non-troublesome dyskinesia, with troublesome dyskinesia), "Off" condition, or asleep. The "On" time without troublesome dyskinesia combined the categories of "On" time without dyskinesia and "On" time with non-troublesome dyskinesia. The PD Home Diary was collected at both the cDBS Baseline and aDBS Evaluation Phases. The threshold was determined using the hours of "On" time without troublesome dyskinesia for aDBS is no worse than 2 hours per day less than cDBS. The proportion of aDBS subjects exceeding the threshold was the primary endpoint.
Time Frame: About one month
Population: As pre-specified, the analysis population included only Primary Cohort subjects, following the intention-to-treat principle, who initiated the aDBS Evaluation Phase (including both randomized crossover subjects and one mode subjects). Analysis of the primary endpoint is based on the aDBS mode (Single or Dual Threshold) by pooling subjects from randomized crossover and one mode arms. As pre-specified, Directional Stimulation Cohort was not included in the primary objective analysis.
Measure: Number (97.5% Confidence Interval); unit: percentage of participant
Groups:
- Primary Cohort aDBS Single Threshold: Adaptive DBS Single Threshold Mode
  Adaptive DBS: Subjects for whom both aDBS modes are acceptable will receive Dual and Single Threshold aDBS
- Primary Cohort aDBS Dual Threshold: Adaptive DBS DualThreshold Mode
  Adaptive DBS: Subjects for whom both aDBS modes are acceptable will receive Dual and Single Threshold aDBS
Arm/Group | Primary Cohort aDBS Single Threshold | Primary Cohort aDBS Dual Threshold
Number analyzed (Participants) | 35 | 40
percentage of participant | 78.9 [59.4 to NA] — Pre-specified hypothesis testing was one-sided, the lower bound of the 97.5% confidence limit was determined using the MI Clopper-Pearson mean success approach, the upper bound was not calculated. So only the confidence interval lower bound is provided, the upper bound is NA. | 91 [75.6 to NA] — Pre-specified hypothesis testing was one-sided, the lower bound of the 97.5% confidence limit was determined using the MI Clopper-Pearson mean success approach, the upper bound was not calculated. So only the confidence interval lower bound is provided, the upper bound is NA.
Statistical Analysis 1: Comparison: Primary Cohort aDBS Single Threshold; Null Hypothesis: The proportion of subjects with "On" time without troublesome dyskinesia during aDBS single threshold mode Evaluation Period exceeding threshold <= 50%; Alternative Hypothesis: The proportion of subjects with "On" time without troublesome dyskinesia during aDBS single threshold mode Evaluation Period exceeding threshold > 50%; Test type: Superiority; Proportion expressed as a percentage = 78.9, 97.5% CI 1-sided [lower limit 59.4] — The confidence interval lower limit was above the performance goal of 50%, the primary objective was met
Statistical Analysis 2: Comparison: Primary Cohort aDBS Dual Threshold; Null Hypothesis: The proportion of subjects with "On" time without troublesome dyskinesia during aDBS dual threshold mode Evaluation Period exceeding threshold <= 50%; Alternative Hypothesis: The proportion of subjects with "On" time without troublesome dyskinesia during aDBS dual threshold mode Evaluation Period exceeding threshold > 50%; Test type: Superiority; Proportion expressed as a percentage = 91.0, 97.5% CI 1-sided [lower limit 75.6] — The confidence interval lower limit was above the performance goal of 50%, the primary objective was met

2. Secondary Outcome: Stimulation Energy Use
Description: Total electrical energy delivered (TEED) for aDBS as compared with cDBS, calculated as TEED at aDBS - TEED at cDBS.
Time Frame: About one month
Population: As pre-specified, the analysis population included only Primary Cohort subjects, following the intention-to-treat principle, who initiated the aDBS Evaluation Phase (including both randomized crossover subjects and one mode subjects). Analysis of the primary endpoint is based on the aDBS mode (Single or Dual Threshold) by pooling subjects from randomized crossover and one mode arms. As pre-specified, Directional Stimulation Cohort was not included in the secondary objective analysis.
Measure: Mean (97.5% Confidence Interval); unit: micro Watts
Groups:
- aDBS Dual Threshold: Adaptive DBS DualThreshold Mode
  Adaptive DBS: Subjects for whom both aDBS modes are acceptable will receive Dual and Single Threshold aDBS
Arm/Group | aDBS Single Threshold | aDBS Dual Threshold
Number analyzed (Participants) | 35 | 40
micro Watts | -22.3 [-42.0 to -2.6] | -22.3 [-48 to 3.3]
Statistical Analysis 1: Comparison: aDBS Single Threshold; Null Hypothesis: Mean Difference between aDBS single threshold (Evaluation Phase) minus cDBS (Baseline Phase) for TEED >= 0; Alternative Hypothesis: Mean Difference between aDBS single threshold (Evaluation Phase) minus cDBS (Baseline Phase) for TEED < 0; Test type: Superiority; p = 0.0120, t-test, 2 sided — Nominal p-value is provided
Statistical Analysis 2: Comparison: aDBS Dual Threshold; Null Hypothesis: Mean Difference between aDBS dual threshold (Evaluation Phase) minus cDBS (Baseline Phase) for TEED >= 0; Alternative Hypothesis: Mean Difference between aDBS dual threshold (Evaluation Phase) minus cDBS (Baseline Phase) for TEED < 0; Test type: Superiority; p = 0.0491, t-test, 2 sided — Nominal p-value is provided

3. Other Pre Specified Outcome: Safety (Stimulation-related AEs)
Description: To characterize stimulation-related adverse events
Time Frame: About one month
Population: As pre-specified, the analysis population included only Primary Cohort subjects, following the intention-to-treat principle, who initiated the aDBS Evaluation Phase (including both randomized crossover subjects and one mode subjects). Analysis of the primary endpoint is based on the aDBS mode (Single or Dual Threshold) by pooling subjects from randomized crossover and one mode arms. As pre-specified, Directional Stimulation Cohort was not included in the analysis of this objective.
Measure: Count of Participants; unit: Participants
Groups:
- Primary Cohort at cDBS Baseline: Subjects who were included in the Full Analysis Set during cDBS Baseline
- Primary Cohort: aDBS Single Threshold Mode: Adaptive DBS Single Threshold Mode, including subjects in Full Analysis Set who were either randomized to crossover periods or received one mode
- Primary Cohort: aDBS Dual Threshold Mode: Adaptive DBS Dual Threshold Mode, including subjects in Full Analysis Set who were either randomized to crossover periods or received one mode
Arm/Group | Primary Cohort at cDBS Baseline | Primary Cohort: aDBS Single Threshold Mode | Primary Cohort: aDBS Dual Threshold Mode
Number analyzed (Participants) | 45 | 35 | 40
Participants | 3 | 8 | 5

ADVERSE EVENTS:
Time Frame: From subject enrollment to subject last visit or subject exit, an average of 15 months.
Description: In order to assess the adverse events by intervention/mode, adverse events that were related to device and/or therapy, i.e., stimulation related adverse events are presented here. The groups are: Enrollment to Randomization, PC aDBS Single Mode, PC aDBS Dual Mode, DS aDBS Single Mode, DS aDBS Dual Mode. Subjects may be in more than one group. Enrollment to Randomization includes cDBS and aDBS setup and adjustment phases. One death was not related to device, procedure, therapy, or stimulation.
Groups:
- Enrollment to Randomization: Included the adverse events occurred from enrollment to randomization where subjects were either under cDBS or temporarily under aDBS during setup and adjustment phase. This group included subjects from both Primary Cohort and Directional stimulation Cohort.
- Primary Cohort aDBS Single Threshold Mode: Included the adverse events occurred after Primary Cohort subjects entered the aDBS Evaluation Phase. This group combined the subjects from the crossover arm and one mode arm where the adverse events happened during the aDBS Single Threshold Mode.
- Primary Cohort aDBS Dual Threshold Mode: Included the adverse events occurred after Primary Cohort subjects entered the aDBS Evaluation Phase. This group combined the subjects from the crossover arm and one mode arm where the adverse events happened during the aDBS Dual Threshold Mode.
- Directional Stimulation Cohort aDBS Single Threshold Mode: Included the adverse events occurred after Directional Stimulation Cohort subjects entered the aDBS Evaluation Phase. This group combined the subjects from the crossover arm and one mode arm where the adverse events happened during the aDBS Single Threshold Mode.
- Directional Stimulation Cohort aDBS Dual Threshold Mode: Included the adverse events occurred after Directional Stimulation Cohort subjects entered the aDBS Evaluation Phase. This group combined the subjects from the crossover arm and one mode arm where the adverse events happened during the aDBS Dual Threshold Mode.
Arm/Group | Enrollment to Randomization | Primary Cohort aDBS Single Threshold Mode | Primary Cohort aDBS Dual Threshold Mode | Directional Stimulation Cohort aDBS Single Threshold Mode | Directional Stimulation Cohort aDBS Dual Threshold Mode
All-Cause Mortality (participants affected / at risk) | 0/85 | 1/35 | 0/40 | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/85 | 1/35 | 0/40 | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 32/85 | 10/35 | 16/40 | 4/13 | 5/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrollment to Randomization (N=85) | Primary Cohort aDBS Single Threshold Mode (N=35) | Primary Cohort aDBS Dual Threshold Mode (N=40) | Directional Stimulation Cohort aDBS Single Threshold Mode (N=13) | Directional Stimulation Cohort aDBS Dual Threshold Mode (N=15)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrollment to Randomization (N=85) | Primary Cohort aDBS Single Threshold Mode (N=35) | Primary Cohort aDBS Dual Threshold Mode (N=40) | Directional Stimulation Cohort aDBS Single Threshold Mode (N=13) | Directional Stimulation Cohort aDBS Dual Threshold Mode (N=15)
Gait disturbance (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Propulsive gait (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 16 (22) | 3 (4) | 4 (5) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 1 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Freezing phenomenon (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Parkinson's disease (worsening) (Nervous system disorders) | 13 (14) | 5 (6) | 8 (9) | 2 (2) | 3 (4)
Tremor (Nervous system disorders) | 7 (8) | 3 (3) | 1 (1) | 2 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT04547712/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT04547712/SAP_001.pdf